CLINICAL TRIAL: NCT03847090
Title: Establishing the Safety and Efficacy of Reloxaliase (Oxalate Decarboxylase) in Patients With Enteric Hyperoxaluria: A Phase III Randomized, Double-Blind, Placebo-Controlled Study (URIROX-2)
Brief Title: Establishing the Safety and Efficacy of Reloxaliase in Patients With Enteric Hyperoxaluria
Acronym: URIROX-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim Analysis -
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLN-177-302; 2018-000921-29 (EudraCT Number)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Enteric Hyperoxaluria
Keywords: kidney stone; hyperoxaluria; enteric hyperoxaluria; oxalate; kidney calcification
MeSH Terms: conditions — Kidney Calculi; Hyperoxaluria | interventions — reloxaliase; oxalate decarboxylase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reloxaliase (Experimental): Reloxaliase (ALLN-177) 142 mg of oxalate decarboxylase (equivalent to 3,750 units of enzyme activity) per capsule
  Interventions: Drug: Reloxaliase
- placebo (Placebo Comparator): placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reloxaliase — Reloxaliase 2 capsules, orally, with each meal/snack, 3 to 5 times per day
  Other Names: ALLN-177; Oxalate decarboxylase
  Arms: Reloxaliase
Drug: Placebo — Placebo 2 capsules, orally, with each meal/snack, 3 to 5 times per day
  Other Names: Placebo capsule
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the efficacy, durability and long-term safety of reloxaliase in patients with enteric hyperoxaluria.

DETAILED DESCRIPTION:
This is a phase 3, global, multi-center, randomized, double-blind, placebo-controlled study. This study is designed to determine the short- and long-term efficacy of reloxaliase in terms of reducing urinary oxalate excretion and clinical benefits compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent
2. Age 18 years or older
3. Has an underlying enteric disorder associated with malabsorption with known or suspected history of hyperoxaluria (e.g., history of kidney stones or oxalate nephropathy)
4. Urinary oxalate ≥ 50 mg/24 hr
5. Has at least 1 documented kidney stone within 2 years

Exclusion Criteria:

1. Acute renal failure or estimated glomerular filtration rate (eGFR) < 30 mL/minute/1.73 m2
2. Has a known genetic, congenital, or other cause of kidney stones
3. Unable or unwilling to discontinue Vitamin C supplementation >200mg daily
4. Cannot establish baseline kidney stone burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in 24-hour urinary oxalate excretion during Weeks 1 to 4 | 4 weeks
  Efficacy will be assessed based on percent change from baseline to the average across Weeks 1 to 4, derived from all 24-hour collections during Weeks 1 to 4 on treatment
Proportion of subjects with kidney stone disease progression (composite of symptomatic kidney stone(s) or finding of new or enlarged kidney stone(s) on imaging) | up to 48 months
  Efficacy will be assessed by comparing kidney stone disease progression event rate on reloxaliase vs. placebo

SECONDARY OUTCOMES:
Percent change from baseline in 24-hour urinary oxalate excretion during Weeks 16-24 | 24 weeks
  Efficacy will be assessed based on percent change from baseline to the average across Weeks 16-24, derived from all 24-hour collections during Weeks 16-24 on treatment
Proportion of subjects with a ≥ 20% reduction from baseline in 24-hour urinary oxalate excretion during Weeks 1-4 | 4 weeks
  Efficacy will be assessed based on proportion of subjects with ≥ 20% reduction from baseline to the average across Weeks 1-4, derived from all 24-hour collections during Weeks 1-4 on treatment
Hospitalizations or emergency room (ER) visits or procedures for the management of kidney stones | up to 48 months
  Efficacy will be assessed by comparing utilization on reloxaliase vs. placebo
Change in estimated glomerular filtration rate (eGFR) from baseline | up to 48 months
  Efficacy will be assessed by comparing the rate of change in eGFR on reloxaliase vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Clark, MD, Study Director — Allena Pharmaceuticals Inc
Locations (113):
- United States (64):
  - University of Alabama- Department of Urology, Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Aventiv Research Inc., Mesa, Arizona
  - Arizona Kidney Disease and Hypertension Center (AKDHC)- Phoenix, Peoria, Arizona
  - Arizona Kidney Disease and Hypertension Center (AKDHC)- Glendale, Phoenix, Arizona
  - Mayo Mercy Hospital, Phoenix, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Renal Consultants Medical Group, Granada Hills, California
  - Amicis Research, Northridge, California
  - University of California, San Diego (UCSD) Health System, San Diego, California
  - University of California- San Francisco (UCSF), San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Sutter Health- Sacramento, Vacaville, California
  - Yale University School of Medicine, New Haven, Connecticut
  - South Florida Nephrology Group PA Research Div, Coral Springs, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Quantum Clinical Research, Hialeah, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Pro-Care Research Center, Corp, Miami Gardens, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Idaho Catalyst Clinical Research, Idaho Falls, Idaho
  - Idaho Urologic Institute, Meridian, Idaho
  - IU Health Physicians, Carmel, Indiana
  - Indiana University (IU) Nephrology, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Associates, LLC d/b/a/ Chesapeake Urology Research Associates, Glen Burnie, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic- Department of Nephrology Hyperoxaluria Center, Rochester, Minnesota
  - University of Missouri Healthcare, Columbia, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - Sheldon J. Freedman, MD, Las Vegas, Nevada
  - New York Presbyterian/Queens, Flushing, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - New York University School of Medicine- Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina (UNC) - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - University of Cincinnati (UC) - Department of Nephrologyv, Cincinnati, Ohio
  - Ohio State University (OSU)-Renal Division, Columbus, Ohio
  - Clinical Research Solutions- Middleburg Heights, Middleburg Heights, Ohio
  - Genito-Urinary Surgeons, Toledo, Ohio
  - Oregon Health and Science University (OHSU), Portland, Oregon
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Lifespan Physician Group Minimally Invasive Urology Institute, Providence, Rhode Island
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Accelemed Research Institute, Austin, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Baylor Scott and White Research Institute- Temple, Temple, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - University of Wisconsin - Division of Nephrology, Madison, Wisconsin
- Medizinische Universitat Wien, Innere Medizin III, Vienna, Austria
- Belgium (3):
  - UVC Brugmann University Hospital- Centre Hospitalier Universitaire, Brussels
  - Universite Libre de Bruxelles -Hospital Erasme, Brussels
  - University Hospital Gent, Ghent
- Brazil (4):
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da UFMG, Belo Horizonte
  - Faculdade de Medicina do ABC, Santo André
  - Pesquisare Saude, Santo André
- Canada (4):
  - University of Alberta- Division of Urology, Edmonton, Alberta
  - Silverado Research Inc, Victoria, British Columbia
  - Centre de Recherche Du Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
- Polyclinic Solme, Zagreb, Croatia
- France (4):
  - Hopital Beaujon_AP_HP, Clichy
  - AP-HM Hospital de la Conception, Marseille
  - Hospital Tenon-AP-HP, Paris
  - CHRU de Nancy-Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (2):
  - Charite Universitaetsmedizin- Berlin, Berlin
  - Klinikum der Universitaet- Muenche, München
- Italy (3):
  - Azienda USL Toscana Centro-Ospedale Santa Maria Nuova, Florence
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST, Genova
  - Fondazione Policlinico Universitario A.Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
- Mexico (4):
  - Invesclinic MX, Irapuato, Gto, C.P
  - ICARO Investigaciones en Medicina SA de CV/Hospital Christus Muguerza, Chihuahua City
  - Clinstile, S.A. de C.V- Col. Roma Norte Delegacion, Cuauhtémoc
  - Centro specializado en Diabetes, Obesidad y Prevencion de Enfermedades Cardiovasculares, Mexico City
- Portugal (2):
  - Hospital Fernando da Fonseca, Amadora
  - Centro Hospitalar Universitario de Sao Joao, Porto
- Romania (5):
  - Sana Medical Center, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Universitar de Urgenta Bucuresti, Bucharest
  - ClinTrial/County Hospital Caracal, Caracal
  - Centru de Diagnostic si Tratament Affidea- Medicina Interna, Constanța
- Russia (6):
  - Clinic of Urology LLC, Penza
  - LLC Medsi St Petersburg, Saint Petersburg
  - S.M Kirov Military Medical Academy, Saint Petersburg
  - Medical Center "Reavita Med StP" LLC, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - Saratov State Medical University, n.a. V.I. Razumosky, Saratov
- Spain (3):
  - Fundacio Puigvert, Barcelona
  - Hospital Universitari de Girona, Girona
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (2):
  - Inselspital, Universitaetsspital Bern Inselspital Bern University Hospital, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV) Lausanne Nephrology Department, Lausanne
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - Darent Valley Hospital, Dartford
  - The Royal Free Hospital, London
  - South Tyneside District Hospital - South Shields, South Shields
  - Wrexham Maelor Hospital, Wrexham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langman CB, Grujic D, Pease RM, Easter L, Nezzer J, Margolin A, Brettman L. A Double-Blind, Placebo Controlled, Randomized Phase 1 Cross-Over Study with ALLN-177, an Orally Administered Oxalate Degrading Enzyme. Am J Nephrol. 2016;44(2):150-8. doi: 10.1159/000448766. Epub 2016 Aug 17. PMID 27529510
- [Background] Lingeman JE, Pareek G, Easter L, Pease R, Grujic D, Brettman L, Langman CB. ALLN-177, oral enzyme therapy for hyperoxaluria. Int Urol Nephrol. 2019 Apr;51(4):601-608. doi: 10.1007/s11255-019-02098-1. Epub 2019 Feb 19. PMID 30783888
- See also: A Double-Blind, Placebo Controlled, Randomized Phase 1 Cross-Over Study with ALLN-177, an Orally Administered Oxalate Degrading Enzyme — https://www.ncbi.nlm.nih.gov/pubmed/27529510
- See also: ALLN-177, oral enzyme therapy for hyperoxaluria — https://www.ncbi.nlm.nih.gov/pubmed/30783888